CLINICAL TRIAL: NCT00390117
Title: A Phase I Study of AT7519M Given Twice Weekly in Patients With Advanced Incurable Malignancy
Brief Title: AT7519M in Treating Patients With Advanced or Metastatic Solid Tumors or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I177; CAN-NCIC-IND177 (Registry Identifier: NCI US - Physician Data Query); CDR0000507621 (Other: PDQ)
Record Dates: First submitted 2006-10-18; First posted 2006-10-19 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2020-04

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; Waldenstrom macroglobulinemia; recurrent adult grade III lymphomatoid granulomatosis; adult nasal type extranodal NK/T-cell lymphoma; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Extranodal NK-T-Cell | interventions — 4-(2,6-dichlorobenzoylamino)-1H-pyrazole-3-carboxylic acid piperidin-4-ylamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CDKI AT7519 (Experimental): AT7519M (1 hour IV) on days 1, 4, 8 and 11 every 5 weeks.
  Interventions: Drug: CDKI AT7519; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: CDKI AT7519 — AT7519M (1 hour IV) on days 1, 4, 8 and 11 every 5 weeks.
Other: laboratory biomarker analysis — Pharmacokinetic bioanalysis of the AT7519 plasma concentration data will be performed by BioDynamics Northhampton, U.K. The pharmacokinetic parameters for AT7519 will be determined by Astex Therapeutics as data permits.

SUMMARY:
RATIONALE: AT7519M may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I trial is studying the side effects and best dose of AT7519M in treating patients with advanced or metastatic solid tumors or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the recommended phase II dose of AT7519M in patients with advanced or metastatic solid tumors or refractory non-Hodgkin's lymphoma.
* Determine the safety, tolerability, toxicity profile, and dose-limiting toxicities of this drug in these patients.
* Determine the pharmacokinetic profile of this drug in these patients.
* Correlate the toxicity profile with pharmacokinetics of this drug in these patients.

Secondary

* Assess, preliminarily, the antitumor activity of this drug in these patients.

OUTLINE: This is an open-label, dose-escalation, multicenter study.

Patients receive AT7519M IV over 1-3 hours on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of AT7519M until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity during course 1. Once the MTD has been determined, up to 8 additional patients are treated at the MTD.

Patients undergo blood collection periodically for pharmacokinetic studies. Patients treated at the MTD also undergo tumor tissue biopsies or aspirates and blood collection periodically for additional pharmacodynamic and correlative biomarker studies.

After completion of study therapy, patients are followed at 4 weeks. Patients with complete response, partial response, or stable disease are followed every 3 months thereafter until relapse.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed diagnosis of 1 of the following:

  * Advanced and/or metastatic solid tumor

    * No more than 3 prior regimens for metastatic disease
  * Refractory non-Hodgkin's lymphoma
* Clinically or radiologically documented disease

  * Patients whose only evidence of disease is tumor marker elevation are not eligible
* No untreated brain or meningeal metastases

  * Patients with radiologic or clinical evidence of stable, treated brain metastases are eligible provided they are asymptomatic AND have no requirement for corticosteroids

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 1.25 times upper limit of normal (ULN) OR creatinine clearance ≥ 50 mL/min
* Bilirubin normal
* ALT and AST ≤ 2 times ULN (5 times ULN if patient has documented liver metastases)
* Potassium normal
* Calcium normal
* Creatine kinase (CK or CPK) ≤ 2 times ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No pre-existing cardiovascular conditions and/or symptomatic cardiac dysfunction, including any of the following:

  * Significant cardiac event (including symptomatic heart failure or angina) within the past 3 months or any cardiac disease that, in the opinion of the investigator, increases the risk for ventricular arrhythmia
  * Any history of ventricular arrhythmia, which was symptomatic or required treatment (CTC grade 3), including multifocal PVCs, bigeminy, trigeminy, or ventricular tachycardia
  * Uncontrolled hypertension
  * Previous history of QT prolongation with other medication
  * Congenital long QT syndrome
  * QT and QTc, with Bazett's correction, unmeasurable or ≥ 460 msec on screening ECG
  * LVEF < 45 % by MUGA for patients with significant cardiac history (i.e., myocardial infarction, severe hypertension, or arrhythmia) or prior doxorubicin (> 450 mg/m²)
* No active or uncontrolled infections
* No serious illness or medical condition that would preclude study compliance
* No peripheral neuropathy > grade 1

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 21 days since prior cytotoxic chemotherapy and recovered (solid tumors)
* At least 21 days since prior palliative radiotherapy and recovered

  * Exceptions may be made for low-dose, nonmyelosuppressive radiotherapy
* Prior hormonal, immunologic, biologic, or signal transduction inhibitor therapy allowed
* At least 14 days since prior major surgery and recovered (no nonhealing wounds)
* At least 4 weeks since prior steroids
* No other concurrent medications which affect QT/QTc and cannot be discontinued
* No other concurrent experimental drugs or anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-01-05 (Actual); Primary Completion 2012-03-13 (Actual); Study Completion 2013-01-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose as assessed by NCI CTCAE v.30 | from time of 1st dose
Safety, tolerability, toxicity profile, and dose-limiting toxicities as assessed by NCI CTCAE v.30 | from time of 1st dose
Pharmacokinetic profile as measured on days 1, 2, and 4 in course 1 | one month
  during cycle 1
Correlation of toxicity profile with pharmacokinetics | after completion of each dose level

SECONDARY OUTCOMES:
Preliminary antitumor activity of treatment in patients with measurable disease | Every 60 days
  after every second cycle
Overall response (complete and partial response) rate | Every 60 days
  after every second cycle
Response duration (median and range) | after progression

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Hotte, MD, Study Chair — Margaret and Charles Juravinski Cancer Centre; Eric X. Chen, MD, PhD, Study Chair — Princess Margaret Hospital, Canada
Locations (2):
- Canada (2):
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Univ. Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chen EX, Hotte S, Hirte H, Siu LL, Lyons J, Squires M, Lovell S, Turner S, McIntosh L, Seymour L. A Phase I study of cyclin-dependent kinase inhibitor, AT7519, in patients with advanced cancer: NCIC Clinical Trials Group IND 177. Br J Cancer. 2014 Dec 9;111(12):2262-7. doi: 10.1038/bjc.2014.565. Epub 2014 Nov 13. PMID 25393368
- [Derived] Malumbres M, Barbacid M. Cell cycle, CDKs and cancer: a changing paradigm. Nat Rev Cancer. 2009 Mar;9(3):153-66. doi: 10.1038/nrc2602. PMID 19238148